CLINICAL TRIAL: NCT05069181
Title: Pilates Mat Versus Cervical Stabilization Exercises on Myoelectric Activity of Cervical Muscles, Craniovertebral Angle, Pain and Function in Young Adults With Forward Head Posture: Randomized Controlled Trial
Brief Title: Pilates Mat Versus Cervical Stabilization Exercises on Myoelectric Activity of Cervical Muscles in Forward Head Posture
Acronym: FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, Doctor of physical therapy, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/003349
Record Dates: First submitted 2021-09-16; First posted 2021-10-06 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Diseases
Keywords: Forward head posture; Craniovertebral angle; Pilates mat exercises
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates mat exercises (Experimental): one hour Pilates exercises with 10 min warm up and 5-10 min cooling down
  Interventions: Other: Pilates mat exercises; Other: conventional physiotherapy
- cervical stabilization exercises (Experimental): training of deep cervical flexor muscles with pressure biofeedback unit
  Interventions: Other: cervical stabilization exercises; Other: conventional physiotherapy
- conventional physiotherapy (Active Comparator): 10 min hot pack on cervical area range of motion exercises and isometric neck exercises as a home program
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Pilates mat exercises — Pilates mat exercises: Each Pilates session will last for one hour and commence with a 10 minute warm up and finish with a 10 min cool down. The subjects will be taught the 5 key elements of Pilates (lateral costal breathing, centring which is a neutral position of the lumbar spine with activation of the core muscles, ribcage placement, shoulder blade placement and neutral position of the cervical spine with slight upper cervical flexion at the cranio-cervical junction).
  Pilates exercise program will consist of warm up exercises, main treatment program (10 level) and cooling down exercises.
  Arms: Pilates mat exercises
Other: cervical stabilization exercises — training of deep cervical flexor muscles with pressure biofeedback unit, 20 min/day, 3 days/week for 12 weeks.
  Arms: cervical stabilization exercises
Other: conventional physiotherapy — 10 min hot pack on cervical area range of motion exercises and isometric neck exercises as a home program 3 days/week for 12 weeks

SUMMARY:
see if there is no statistical significant difference between the effects of Pilates mat versus cervical stabilization exercises on myoelectric activity of cervical muscles in young adults with forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) increases extension of the atlanto-occipital joint and the upper cervical vertebrae as well as flexion of the lower cervical and upper thoracic vertebrae. Furthermore, this posture causes persistent and abnormal contraction of the suboccipital, neck, and shoulder muscles. Additionally, the muscles around the head and shoulders, including the trapezius, sternocleidomastoid, suboccipital, and temporal, are affected by FHP, which further worsens postural deformity. FHP is the most common deviation from ideal head posture and is characterized by the head projecting forward into the sagittal plane such that it is anterior to the trunk. Head in forward posture can add up to thirty pounds of abnormal leverage on the cervical spine, which pull the entire spine out of alignment, in addition, loss of the physiological lordosis could be a possible cause of pain due to muscular imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders aged 18-25 years old with forward head posture will be included in this study
* Subjects have forward head posture if craniovertebral angle ≤ 50.
* Subjects complain non- specific neck pain for at least 3 months or at least two episodes of non-specific neck pain during the last three months.
* Normal body mass index

Exclusion Criteria:

* Subjects with any spinal problems
* Subjects with experience in Pilates exercises through the last 3 months of the start of intervention will be excluded from the study
* Previous surgery in the neck and shoulder regions
* Current participation in a structured exercises program
* Neurological symptoms of the upper extremities during screening tests (e.g., Spurling test and upper limb tension tests)
* Red flags suggesting of cancer, infection, vascular insufficiency
* Cervical radiculopathy or myelopathy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Myoelectric activity of cervical muscles | up to twelve weeks
  by surface electromyography (EMG)
Craniocervical angle | up to twelve weeks
  by photogrammetric method.

SECONDARY OUTCOMES:
Pain intensity of neck area | up to twelve weeks
  by visual analogue scale 10 cm line with 2 ends, 0 and 10 ends 0 end means no pain 10 end means the worst pain
function of daily life | up to twelve weeks
  by neck disability index

CONTACTS AND LOCATIONS:
Overall Officials: Haytham M Elhafez, Professor, Study Director — professor of physical therapy- cairo university
Locations (1):
- Faculty of Physical Therapy-Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we will share the results of the trial 1-craniovertebral angle 2-myoelevtric activity of cervical muscles 3-pain of neck area 4-function and neck disability
Supporting Information: Study Protocol
Time Frame: one year
Access Criteria: the criteria will be accessed by the publication of trials in international journal